CLINICAL TRIAL: NCT00087932
Title: Socioeconomic Diversity of CAM Integration in Oncology
Brief Title: Socioeconomic Influences on Complementary and Alternative Medicine Use in Cancer Treatment
Status: Completed | Type: Observational
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Other Study IDs: R21AT000880 (NIH)
Record Dates: First submitted 2004-07-15; First posted 2004-07-16 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Neoplasms
Keywords: Complementary Therapies
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to determine whether differences in the use of complementary and alternative medicine (CAM) are influenced by the socioeconomic status and ethnicity of cancer patients.

DETAILED DESCRIPTION:
The use of CAM is common among patients with cancer. However, there may be differences in participation, treatment preferences, and quality of life that are influenced by socioeconomic factors and ethnicity. This study will compare two distinct socioeconomic groups to determine differences in CAM use.

Participants in this study will complete a questionnaire regarding demographics, socioeconomic status, disease specifics, and facilitators and barriers to CAM use. Participation in an introductory seminar and in various CAM programs will be monitored. Participants will also complete a quality of life scale that will provide insight into the way different populations perceive and use CAM and will identify potential obstacles to integrating CAM into other cancer treatment programs.

ELIGIBILITY:
Inclusion Criteria:

* Cancer diagnosis
* Able to read and understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2001-09; Study Completion 2003-08

CONTACTS AND LOCATIONS:
Overall Officials: June L. Chan, MD, Principal Investigator — University of Michigan
Locations (1):
- Assarian Cancer Center, Novi, Michigan, United States